CLINICAL TRIAL: NCT02980900
Title: The Effect of Protein Ingestion on the Recovery of Skeletal Muscle Function Following Eccentric Exercise.
Acronym: SPADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 181739
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo supplement (Placebo Comparator): Post exercise placebo supplement Pre bed placebo supplement
  Interventions: Dietary Supplement: Post exercise placebo supplement; Dietary Supplement: Pre bed placebo supplement
- Post exercise supplement (Active Comparator): Post exercise protein-polyphenol supplement Pre bed placebo supplement
  Interventions: Dietary Supplement: Post exercise protein-polyphenol supplement; Dietary Supplement: Pre bed placebo supplement
- Pre bed supplement (Active Comparator): Post exercise placebo supplement Pre bed protein-polyphenol supplement
  Interventions: Dietary Supplement: Post exercise placebo supplement; Dietary Supplement: Pre bed protein-polyphenol supplement
- Post exercise + pre bed supplement (Active Comparator): Post exercise protein-polyphenol supplement Pre bed protein-polyphenol supplement
  Interventions: Dietary Supplement: Post exercise protein-polyphenol supplement; Dietary Supplement: Pre bed protein-polyphenol supplement

INTERVENTIONS:
Dietary Supplement: Post exercise protein-polyphenol supplement — Participants will ingest a post exercise protein-polyphenol supplement. This will begin 6 days before eccentric exercise and will end 6 days after eccentric exercise.
  Arms: Post exercise + pre bed supplement; Post exercise supplement
Dietary Supplement: Post exercise placebo supplement — Participants will ingest an isocaloric placebo supplement after exercise. This will begin 6 days before eccentric exercise and will end 6 days after eccentric exercise.
  Arms: Placebo supplement; Pre bed supplement
Dietary Supplement: Pre bed protein-polyphenol supplement — Participants will ingest a protein-polyphenol supplement before bed. This will begin 6 days before eccentric exercise and will end 6 days after eccentric exercise.
  Arms: Post exercise + pre bed supplement; Pre bed supplement
Dietary Supplement: Pre bed placebo supplement — Participants will ingest an isocaloric placebo supplement before bed. This will begin 6 days before eccentric exercise and will end 6 days after eccentric exercise.
  Arms: Placebo supplement; Post exercise supplement

SUMMARY:
The present study will assess the effect of the type and timing of protein ingestion 6 days prior to, and 7 days following eccentric exercise on the time course of 1) the recovery of muscle function, 2) the recovery of perceived muscle soreness, 3) muscle metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are generally healthy and recreationally active

Exclusion Criteria:

* Active cardiovascular disease or hypertension
* Diagnosed metabolic impairment
* Use of nutritional supplements
* Use of anti-inflammatory medications
* Habitual dietary protein intake of <0.8g/kg/day
* Musculoskeletal disorders

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Isokinetic force production of the knee extensor muscles | 14 days

SECONDARY OUTCOMES:
Muscle protein synthesis | 14 days
Thigh volume | 14 days
Perceived muscle soreness | 14 days
Isometric force production of the knee extensor muscles | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sport and Health Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jameson TSO, Pavis GF, Dirks ML, Lee BP, Abdelrahman DR, Murton AJ, Porter C, Alamdari N, Mikus CR, Wall BT, Stephens FB. Reducing NF-kappaB Signaling Nutritionally is Associated with Expedited Recovery of Skeletal Muscle Function After Damage. J Clin Endocrinol Metab. 2021 Jun 16;106(7):2057-2076. doi: 10.1210/clinem/dgab106. PMID 33710344